CLINICAL TRIAL: NCT00338754
Title: A Phase 2/3, Randomized, Double-Blind, Placebo Controlled, Multicenter Study of Efficacy and Safety of Adalimumab in Japanese Subjects With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: Adalimumab in Adult Japanese Subjects With Moderate to Severe Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Collaborators: Eisai Limited (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M04-688
Record Dates: First submitted 2006-06-18; First posted 2006-06-20 (Estimated); Last update posted 2007-09-11 (Estimated); Status verified 2007-09

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

INTERVENTIONS:
Drug: Human anti-TNF monoclonal antibody adalimumab/ up to 24 weeks

SUMMARY:
The purpose of the study is to assess the efficacy and safety of repeated administration of adalimumab in adult Japanese subjects with moderate to severe chronic plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Subject was age 20 or older and in good health (Investigator discretion) with a recent stable medical history.
* Subject had a clinical diagnosis of psoriasis for at least 6 months, and had moderate to severe plaque psoriasis

Exclusion Criteria:

* Subject had previously received anti-TNF therapy.
* Subject cannot discontinue systemic therapies and/or topical therapies for the treatment of psoriasis and cannot avoid UVA, UVB or PUVA phototherapy
* Subject is taking or requires oral or injectable corticosteroids
* Subject considered by the investigator, for any reason, to be an unsuitable candidate for the study
* Female subject who is pregnant or breast-feeding or considering becoming pregnant

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2005-11

PRIMARY OUTCOMES:
Proportion of subjects with clinical response relative to Baseline PASI score

SECONDARY OUTCOMES:
QoLs
Clinical response indicators
Safety parameters

CONTACTS AND LOCATIONS:
Overall Officials: Noritaka Inomata, Ph.D., Study Director — Abbott Japan Co.,Ltd
Locations (8):
- Japan (8):
  - Chugoku
  - Chūbu
  - Hokkaido
  - Kanto
  - Kinki
  - Kyusyu
  - Shikoku
  - Tōhoku